CLINICAL TRIAL: NCT01144715
Title: An Innovative Home Stroke Rehabilitation and Monitoring System
Brief Title: Rehabilitation of the Stroke Hand at Home
Acronym: HAAPI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kinetic Muscles (Industry)
Collaborators: The Cleveland Clinic (Other); Emory University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NS070646; 1RC3NS070646-01 (NIH)
Record Dates: First submitted 2010-06-11; First posted 2010-06-16 (Estimated); Results first posted 2014-11-27 (Estimated); Last update posted 2014-11-27 (Estimated); Status verified 2014-10

CONDITIONS: Stroke
Keywords: Stroke Rehabilitation; Home rehabilitation; robotic therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hand Mentor Therapy (Experimental): Use of the Hand Mentor (TM) Stroke Therapy Device at home for 8 weeks
  Interventions: Device: Hand Mentor (TM) robotic stroke therapy device
- Control (Active Comparator): Self administered home therapy program
  Interventions: Device: Home Therapy Program

INTERVENTIONS:
Device: Hand Mentor (TM) robotic stroke therapy device — The goal of the Hand Mentor ™ (TM) device is to improve Active Range of Motion in the distal musculature of the paretic limb of patients with stroke. Development of HM patient protocols are based on basic principles of motor learning: the protocols actively engage the patient in activities, progressively increase task difficulty based on patient performance, actively assist patient if necessary (i.e. patient is not passive), provide meaningful feedback at regular intervals, require sensorimotor integration and incorporate the use of tasks that that are intended to transfer to distal motor performance.
  Arms: Hand Mentor Therapy
Device: Home Therapy Program — Subjects in the control group will be instructed in a self administered home therapy program
  Arms: Control

SUMMARY:
The purpose of this research is to evaluate a therapy delivery system for stroke patients that provide accessible, affordable stroke care. User-friendly home therapy robots and a telerehabilitation system are combined to monitor and provide therapy that is accessible for patients in rural and underserved locations. The robotic-based home therapy intervention will produce significantly greater improvement in upper extremity motor function than Usual and Customary Care enhanced with a (non-robotic) home therapy upper extremity rehabilitation program at the end of 8 weeks of home therapy.

DETAILED DESCRIPTION:
The primary purpose of this proposal is to evaluate a combined clinic/home robotic-based stroke therapy delivery and monitoring system in rural and underserved locations that provides accessible, effective and affordable care for stroke survivors with residual limb impairment. The study is a prospective, single-blind, multi-site Randomized Controlled Trial. A total of 96 patients within 6 months post-stroke will be enrolled and randomly assigned to one of two groups: robotic based home therapy or a self administered (non-robotic) home therapy program.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ischemic or hemorrhagic stroke
* within 6 months of admission to in-patient rehabilitation
* Persistent hemiparesis
* Proximal Upper Extremity voluntary activity
* Preserved cognitive function
* Difficult access to an organized stroke rehabilitation program

Exclusion Criteria:

* Not independent before stroke
* Hemispatial neglect
* Significant other illnesses

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Alberts, PhD, Principal Investigator — The Cleveland Clinic; Steve L Wolf, PhD, Principal Investigator — Emory University Medical School
Locations (2):
- United States (2):
  - Emory University School of Medicine, Atlanta, Georgia
  - Cleveland Clinic Foujndation, Cleveland, Ohio

REFERENCES:
- [Derived] Linder SM, Rosenfeldt AB, Bay RC, Sahu K, Wolf SL, Alberts JL. Improving Quality of Life and Depression After Stroke Through Telerehabilitation. Am J Occup Ther. 2015 Mar-Apr;69(2):6902290020p1-10. doi: 10.5014/ajot.2015.014498. PMID 26122686
- [Derived] Wolf SL, Sahu K, Bay RC, Buchanan S, Reiss A, Linder S, Rosenfeldt A, Alberts J. The HAAPI (Home Arm Assistance Progression Initiative) Trial: A Novel Robotics Delivery Approach in Stroke Rehabilitation. Neurorehabil Neural Repair. 2015 Nov-Dec;29(10):958-68. doi: 10.1177/1545968315575612. Epub 2015 Mar 17. PMID 25782693
- [Derived] Linder SM, Rosenfeldt AB, Reiss A, Buchanan S, Sahu K, Bay CR, Wolf SL, Alberts JL. The home stroke rehabilitation and monitoring system trial: a randomized controlled trial. Int J Stroke. 2013 Jan;8(1):46-53. doi: 10.1111/j.1747-4949.2012.00971.x. PMID 23280269

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hand Mentor Therapy | Control
Started | 51 | 48
Completed | 47 | 45
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Power analysis to achieve .80 power, alpha=0.05, two-tailed, in differential change across groups in Fugl-Meyer during the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hand Mentor Therapy | Control | Total
Number analyzed (Participants) | 51 | 48 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (12.2) | 59.1 (14.1) | 57.5 (13.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 36 | 74
  >=65 years | 13 | 12 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 31 | 33 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 26 | 48
  White | 28 | 20 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 48 | 48 | 96
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 51 | 48 | 99

OUTCOME MEASURES:

1. Primary Outcome: Action Research Arm Test (ARAT)
Description: The amount of recovery of arm-hand function is measured with the Action Research Arm Test (ARAT). The ARAT assesses activity limitations of the upper extremity. It includes 19 items divided into four subscales: grasp, grip, pinch, and gross movement. Scores range from 0-to-57 with a higher score indicating a better outcome.
Time Frame: End of treatment at 8 weeks post enrolment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hand Mentor Therapy | Control
Number analyzed (Participants) | 51 | 48
units on a scale | 39.47 (19.83) | 39.89 (17.13)

2. Secondary Outcome: Wolf Motor Function Test
Description: The Wolf Motor Function Test (WMFT) is used to measure the degree of function using timed tasks. The WMFT is a 17-item measure used to assess activity limitations of the upper extremity. It is comprised of 2 strength items and 15 timed task performance items. The task performance items begin with the measurement of simple proximal movements and progress to more complex distal and whole limb movements. The WMFT yields two scores: 1) a functional ability score quantifying quality of performance, and 2) a timed score quantifying speed of performance in seconds. A shorter time is better outcome.
Time Frame: End of treatment at 8 weeks post enrolment
Measure: Geometric Mean (Standard Deviation); unit: Seconds
Arm/Group | Hand Mentor Therapy | Control
Number analyzed (Participants) | 51 | 48
Seconds | 8.67 (4.76) | 7.92 (3.97)

3. Secondary Outcome: Fugl-Meyer Upper Extremity Test
Description: Upper Extremity neurological impairment will be measured using the Fugl-Meyer Upper Extremity Test (FMA). The FMA is an impairment-based measure consisting of 33 movements with higher scores indicating increased ability of the patient to move out of synergistic patterns toward more isolated movements. Movement quality of the affected UE is compared to the non-affected UE on 0-2 ordinal scale with 0 indicating no movement at all, 1 indicating partial movement of the affected extremity, and 2 indicating movement equivalent to the non-affected UEs. The score ranges from 0-to-66.
Time Frame: End of Treatment at 8 weeks post enrolment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hand Mentor Therapy | Control
Number analyzed (Participants) | 51 | 48
units on a scale | 43.43 (15.64) | 42.89 (14.58)

4. Secondary Outcome: Stroke Impact Scale (SIS)
Description: Quality of Life changes are measured with the Stroke Impact Scale questionnaire. The SIS is a self-rated QOL questionnaire that addresses several domains following stroke: physical strength, memory, feelings and emotions, communication, activities of daily living (ADL), mobility, hand use, meaningful activities, and overall percentage recovery from the stroke. We report the Hand Function subscale, which ranges from 0-to-100. A higher score reflects better hand function.
Time Frame: End of treatment at 8 weeks post enrolment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hand Mentor Therapy | Control
Number analyzed (Participants) | 51 | 48
units on a scale | 49.4 (33.5) | 57.6 (28.2)

ADVERSE EVENTS:
Arm/Group | Hand Mentor Therapy | Control
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/48
Other Adverse Events (participants affected / at risk) | 6/51 | 5/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hand Mentor Therapy (N=51) | Control (N=48)
Lost balance and fell (General disorders) | 3 (3) | 5 (5) — Lost balance and fell
Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject experienced an ulcer
Recurrent stroke (Vascular disorders) | 1 (1) | 0 (0) — One patient suffered a transient ischemic stroke and was withdrawn from the study.
Depression (Psychiatric disorders) | 1 (1) | 0 (0) — A patient reported that she felt she was regressing, and she was frustrated and depressed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days